CLINICAL TRIAL: NCT05656183
Title: CardioSeq: A Prospective, Single-Center, Open-label Study to Evaluate the Impact of Whole Genome Sequencing (WGS) in Individuals With Cardiovascular Disease
Brief Title: CardioSeq: Impact of WGS in Individuals With CVD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Illumina, Inc. (Industry)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ILMN-007
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): To investigate the diagnostic efficacy of WGS and its impact on clinical management compared to usual care in individuals with cardiovascular disease. Diagnostic yield and changes of management (CoM) will be assessed both within the WGS group and compared to a contemporaneous, matched (2:1) usual care (UC) group sourced from EHR records.
  Interventions: Diagnostic Test: TruGenome Cardiovascular Disease test

INTERVENTIONS:
Diagnostic Test: TruGenome Cardiovascular Disease test — The TruGenome Cardiovascular Disease (CVD) test which consists of an in-silico 200 gene cardiovascular disease panel, a further 4 genes with cardiovascular disease risk alleles, 10 pharmacogenomic genes, 35 non-cardiovascular ACMG secondary finding genes and a polygenic risk score (PRS) for coronary artery disease (CAD) will be utilized in this study.

SUMMARY:
This is a prospective, single-center, open-label study to investigate the diagnostic efficacy of the TruGenome CVD test and its impact on clinical management compared to usual care in individuals with cardiovascular disease. Diagnostic yield and changes of management (CoM) will be assessed both within the WGS group and compared to a contemporaneous, matched (2:1) usual care (UC) group sourced from EHR records.

DETAILED DESCRIPTION:
The TruGenome Cardiovascular Disease (CVD) test which consists of an in-silico 200 gene cardiovascular disease panel, a further 4 genes with cardiovascular disease risk alleles, 10 pharmacogenomic genes, 35 non-cardiovascular ACMG secondary finding genes and a polygenic risk score (PRS) for coronary artery disease (CAD) will be utilized in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥18 years of age
2. Stable ambulatory patients with a cardiology visit within the past year or scheduled within the next 90 days.
3. At least one of the following clinical diagnoses:

   A. Any aortopathy, B. Dyslipidemia, C. Coronary or peripheral arterial disease, D. Heart Failure or cardiomyopathy, E. Any arrythmia
4. Must be able to read, understand, and sign an informed consent

Exclusion Criteria:

1. Individuals with a previously confirmed molecular diagnosis of a known genetic disease with an associated cardiovascular phenotype inclusive of monogenic cardiovascular diseases, chromosomal aneuploidies, and microdeletion disorders.
2. Bone marrow transplant recipients
3. Individuals with severe cognitive dysfunction or diminished capacity who are unable to provide informed consent
4. Patients undergoing active chemotherapy treatment for cancer
5. Patients with end-stage renal disease
6. Patients with poor medical prognosis with a life expectancy <1 year
7. Principal Investigator decides for any reason the study is not in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who receive a new monogenic cardiovascular disease finding | 42 Months
  Quantify the proportion of patients who receive a new monogenic cardiovascular disease finding from the TruGenome CVD test

SECONDARY OUTCOMES:
Number of patients who receive any monogenic cardiovascular disease, cardiovascular risk allele, or cardiovascular pharmacogenomic findings. | 42 Months
  Quantify the proportion of patients who receive monogenic cardiovascular disease, cardiovascular risk allele and/or cardiovascular pharmacogenomic findings.
Number of patients who receive monogenic cardiovascular disease, cardiovascular risk allele, or cardiovascular pharmacogenomic findings leading to a CoM within 3 months (90 days) and 6 months (180 days) after Return of Results (RoR). | Within 3 months (90 days) and 6 months (180 days) after Return of Results
  Quantify the proportion of patients who receive monogenic cardiovascular disease, cardiovascular risk allele, or cardiovascular pharmacogenomic findings leading to a CoM within 3 months (90 days) and 6 months (180 days) after Return of Results (RoR).

OTHER OUTCOMES:
Number of patients who received a CoM (as defined above) compared to a contemporaneous matched (2:1) UC group assessed at patient index date (Return of Results), 3 months (90 days), and 6 months (180 days) thereafter. | Within 3 months (90 days) and 6 months (180 days) after Return of Results
  Quantify the proportion of patients who received a CoM as defined above compared to a contemporaneous matched (2:1) UC group assessed at patient index date (Return of Results), 3 months (90 days), and 6 months (180 days) thereafter.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided